CLINICAL TRIAL: NCT02609854
Title: Sustained Acoustic Medicine for Chronic Low Back Pain Secondary to Herniated Nucleus Pulposus or Other Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP-01
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Low Back Pain (CLBP); Intervertebral Disc Displacement
Keywords: herniated disc; sustained acoustic medicine; ultrasound; CLBP
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Sustained Acoustic Medicine Device (Experimental): Sham Sustained Acoustic Medicine device - the device is to be used 4 hours/day, ≥4 days per week for 8 weeks.
  Interventions: Device: Sham Device
- 3 MHz Sustained Acoustic Medicine Device (Experimental): 3 MHz Sustained Acoustic Medicine device - the device is to be used 4 hours/day, ≥4 days per week for 8 weeks.
  Interventions: Device: Sustained Acoustic Medicine (SAM)

INTERVENTIONS:
Device: Sustained Acoustic Medicine (SAM) — Long-duration, low-intensity therapeutic ultrasound device that is self-applied and wearable, delivering treatment up to 4 hours per day.
  Arms: 3 MHz Sustained Acoustic Medicine Device
Device: Sham Device — Inactive ultrasound device
  Arms: Sham Sustained Acoustic Medicine Device

SUMMARY:
ZetrOZ's Ultrasonic Diathermy device is intended for use as a portable and wearable medical device which, when applied to various areas of the body applies Low Intensity Therapeutic Ultrasound (LITUS) to deep tissues. This device is FDA-cleared for pain reduction, treatment of muscle spasm and joint contracture, and increasing local circulation. This study will look at the use of therapeutic ultrasound to relieve pain and reduce disability in subjects with chronic low back pain, a subset of which will have chronic low back pain due to a herniated disc, over an 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic low back pain, may be secondary to herniated nucleus pulposus (HNP) or other causes
* 18-60 years of age, inclusive
* Has Numeric Rating Scale (NRS) pain severity score of at least 4 for a minimum 5 days over the 1 week Baseline Period prior to being randomized to treatment
* Pain lasting >3 months
* Has MRI from within 2 months prior to Screening (If no recent MRI is available, then subject must agree to have MRI performed prior to randomization of treatment)
* If pain is secondary to HNP: MRI within the last 2 months demonstrating the presence of a herniated disc; herniated disc is laterally located and not centrally located; herniated disc is not sequestered
* Has the presence of radicular pain as assessed by a health care practitioner
* Is willing and able to self-administer treatment daily within their place of residence or during normal daily activity, excluding bathing, showering, or other water activities which may result in submersion of the study device.
* Is maintained on a stable pain management regimen, which may include opioid and/or non-opioid analgesic medications, but must be willing to keep dosage(s) stable through the study period; any dose adjustments that the investigator feels are required during the study period must be discussed with the study sponsor; and the use of any medications must be documented in the subject's Medication Log.
* Be willing to discontinue any other interventional treatment modalities on the lower back during the study period (e.g., transcutaneous electrical nerve stimulation, electronic muscle stimulation, traditional ultrasound).

Exclusion Criteria:

* Cannot successfully demonstrate the ability to put on and take off the device.
* Displays any condition which, in the judgment of the investigator, would make participation in the study unacceptable including, but not limited to, the subject's ability to understand and follow instructions.
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening.
* Has arthritis, bone spurs, stenosis, fusions, or implants near the treatment area.
* Is pregnant.
* Is a prisoner.
* Is non-ambulatory (unable to walk).
* Has a pacemaker.
* Has a malignancy in the treatment area.
* Has an active infection, open sores, or wounds in the treatment area.
* Has impaired sensation in the treatment area, such as caused by chemotherapy or anesthesia.
* Has a known neuropathy (disease of the brain or spinal nerves).
* Has a hereditary disposition (tendency) for excessive bleeding (hemorrhage).
* Has peripheral artery disease.
* Has BMI ≥30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory-Short Form (BPI-SF): Pain Severity | Change from Baseline to Week 8

SECONDARY OUTCOMES:
BPI-SF: Pain Interference | Change from Baseline to Week 8
Oswestry Disability Index | Change from Baseline to Week 8
Numeric Rating Scale: Pain on Flexion | Change from Baseline to Week 8
Numeric Rating Scale: Pain on Extension | Change from Baseline to Week 8

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical Pain Consultants, Dryden, New York
  - Osteopathic Medical Arts, Chapel Hill, North Carolina
  - Weber State University, Ogden, Utah